CLINICAL TRIAL: NCT05609682
Title: The Effect of Gabapentin on Post-Operative Pain in Minimally Invasive Sacrocolpopexy: A Randomized Controlled Pilot Study
Brief Title: Effect of Gabapentin on Post-Operative Pain in Minimally Invasive Sacrocolpopexy
Acronym: GPOP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15207
Record Dates: First submitted 2022-10-03; First posted 2022-11-08 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled pilot trial. Randomization will be computer generated, using a 1:1 allocation and variable block sizes of 2 and 4.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Arm (Placebo Comparator): Standard ERAS protocol post-operative care with placebo
  Interventions: Drug: Placebo
- Gabapentin Arm (Active Comparator): Standard ERAS protocol with scheduled postoperative gabapentin
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — Scheduled gabapentin given for two weeks after surgery
  Arms: Gabapentin Arm
Drug: Placebo — Placebo given for two weeks after surgery
  Arms: Placebo Arm

SUMMARY:
Enhanced recovery after surgery (ERAS) has been synonymous with increasing non-opioid multimodal therapies and decreasing opioid therapies after surgery to improve perioperative care. Gabapentin has been standardized as part of routine adjuvant post-operative enhanced recovery protocols after other surgical specialties surgeries. Limited data is known about the specifics of routine adjuvant post-operative gabapentin in the realm of urogynecology. Sacrocolpopexy has been noted as a highly effective prolapse surgical treatment, especially with apical and multicompartment prolapse. In 2006, approximately 73% of all sacrocolpopexy across the nation are completed through a minimally invasive approach. The role of gabapentin as part of a postoperative pain protocol following minimally invasive sacrocolpopexy (MISC) has yet to be determined.

DETAILED DESCRIPTION:
This will be a randomized controlled pilot trial to determine the effect of a standard postoperative pain protocol with scheduled gabapentin versus placebo in decreasing post-operative pain scores. An institutional review board approach will be obtained and the trial will be registered at Clinicaltrials.gov and the protocol adhered to CONSORT guidelines.

Recruitment will start in October 2022 until completion of pilot study enrollment numbers at OU Health - a single academic center. If patients meet inclusion criteria (see below), willing participants will sign a written consent on their preoperative visit.

Researchers will be recruiting 20 patients per study arm: standard ERAS protocol post-operative care with placebo vs study group given standard ERAS protocol with scheduled postoperative gabapentin for the first two weeks following surgery.

Randomization will be computer generated, using a 1:1 allocation and variable block sizes of 2 and 4. Randomization and packing with opaque bags will be performed by our institution's investigation drug pharmacy. Consents will be signed by trained research assistant(s) and randomization should be maintained throughout the duration of enrollment. Patients will receive their medications concealed within an opaque bag given by the surgical team.

The primary outcome is pain during normal activity and rest via a standardized telephone prompt using the validated surgical pain scale (SPS) on POD 3-5 and 7-10. The SPS uses a numeric range from 0 to 10 with 0 representing no pain and 10 representing the worst pain imaginable. Pain scale will be assessed and opioid consumption will be measured at POD 14-16 during their routine follow up. Patients will be asked the number remaining opiate medications left at their follow up visit.

The secondary outcomes include adverse events, characterized using the National Institute of Health Common Terminology of Criteria for Adverse Events version 5.0. Researchers also plan to collect sociodemographic data: age, parity, race, past medical, and past surgical history. Data from routinely administered validated PFDI-20 and PFIQ-7 forms will also be obtained. Surgical data including concomitant procedures, intra- and perioperative complications, estimated blood loss, length of stay, and whether or not the patient discharges home with a catheter will be noted.

Standard post-operative pain control consists of continuous acetaminophen and/or NSAIDs and as needed oral opiates (oxycodone 5-10mg) for moderate to severe pain. If the patient randomizes to the study group, they will receive 14 days of gabapentin starting on postoperative day (POD) 1. Researchers will utilize a dosing pattern that was previously used in the Wu et al. randomized control trial as it was made in consultation with a geriatric pharmacist. Dosing will include administration of gabapentin 300mg nightly for 3 nights and then be increased to 300mg twice a day for an additional 11 days - a total of 25 tablets. Funding for the study and placebo medications for this study will be provided by an internal grant by the Department of Obstetrics and Gynecology.

Patients will be asked to complete a validated Surgical Pain Scale (SPS) pre-operatively to assess baseline pain. All vaginal and abdominal incisions will be infiltrated with local anesthetic prior to incision for both groups. Both groups will be given a standard senna (8.6mg) with docusate (50mg) daily post-operative bowel regimen as previously published by Patel et al. a.

ELIGIBILITY:
Inclusion Criteria:

• Patients have a diagnosis of uterovaginal prolapse, vaginal vault prolapse, or pelvic organ prolapse (based on International Classification of Diseases [ICD]).

Exclusion Criteria:

* Concurrent sphincter or fistula repair, urethral diverticulectomy or mesh excision
* Current gabapentin or pregabalin use
* Oxygen dependency
* Renal failure or glomerular filtration rate of < 30mL/min
* Daily narcotic usage >2 months - this is to allow us to capture an opiate-naïve patient population to better assess the impact of adjuvant gabapentin

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Examine the efficacy of gabapentin in changing postoperative pain scores | 2 weeks post-op
  Measured using the validated surgical pain scale in which 0 (minimum value) means no pain sensation and 10 (maximum value) means most intense pain imaginable

SECONDARY OUTCOMES:
Post-operative opioid consumption | 2 weeks post-op
  Patients will be asked the number remaining opiate medications left at their follow up visit.
Patient satisfaction | 2 weeks post-op
  Patient satisfaction will be obtained using the Pelvic Floor Disability Index questionnaire in which the symptom scale ranges from 0 = not present to 4 = quite a bit in relation to symptoms and how much they bother the participant.
Degree of somnolence | 2 weeks post-op
  The Pelvic Floor Impact Questionnaire measures how symptoms affect activities, relationships and feelings, ranging from Not at all to Quite a bit.

CONTACTS AND LOCATIONS:
Overall Officials: Lieschen Quiroz, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No